CLINICAL TRIAL: NCT02960061
Title: D2 Radical Resection After Neoadjuvant Chemotherapy Combined With HIPEC for Advanced Gastric Cancer: a Prospective Randomized Controlled Trial
Brief Title: Perioperative Chemotherapy Combined With HIPEC for High-risk Advanced Gastric Cancer
Acronym: HIPEC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPEC-006
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-10

CONDITIONS: Survival
Keywords: Intraperitoneal chemotherapy; gastric cancer; Neo-adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Neoadjuvant Therapy; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIPEC (Experimental): After receiving neoadjuvant chemotherapy and D2 radical resection, Hyperthermic intraperitoneal perfusion chemotherapy is conducted,4 catheters are placed in 4 position in the peritoneal cavity: ① under the left diaphragm ② hepatorenal recess ③ left pelvis ④ right pelvis.catheters, all four tubes are connected to the perfusion device.Perfusion prescription: cycle 1, Paclitaxel 75mg/ m2 diluted with 3000ml normal saline heated up to a fixed temperature of 43°C circulate continuously for 60min at a speed of 400-500ml/h; cycle 2 start within 24-48 hours after cycle 1, dosage of paclitaxel adjust to 100mg/ m2, the rest of the same. A total of two cycle is administered, routine adjuvant chemotherapy using SOX (oxaliplatin plus S-1 capsule)or XELOX regimens follows within 4-6 weeks.
  Interventions: Drug: Neoadjuvant chemotherapy; Procedure: D2 radical resection; Drug: Hyperthermic intraperitoneal perfusion chemotherapy; Drug: Adjuvant chemotherapy
- controlled group (Sham Comparator): After receiving neoadjuvant chemotherapy and D2 radical resection, patients receive peritoneal lavage with 3000ml distilled water.Adjuvant chemotherapy using SOX or XELOX regimens is administered as routine within 4-6 weeks.
  Interventions: Drug: Neoadjuvant chemotherapy; Procedure: D2 radical resection; Drug: Adjuvant chemotherapy

INTERVENTIONS:
Drug: Neoadjuvant chemotherapy — Eligible patients receive 4 cycles of mDOF(docetaxel 50 mg/ m2 day 1 + oxaliplatin 85 mg/ m2 day 2 + fluorouracil 400 mg/ m2 bolus iv followed by 600 mg/ m2 22 hours chronic infusion, day 2/3 + leucovorin 200 mg/ m2, day2/3; repeated every 14 days ).
Procedure: D2 radical resection — Laparotomy or laparoscopic surgery are chosen according to the preference of the surgeon. Either cases, a throughout peritoneal cavity exploration is required to comfirmed the tumor resectability and peritoneal metastasis. A curative D2 resection is performed if achievable.
Drug: Hyperthermic intraperitoneal perfusion chemotherapy — Two cycle of hyperthermic intraperitoneal perfusion chemotherapy is administered to patients who have received neoadjuvant chemotherapy and D2 resection, dosage and the relative parameter setting is described above.
  Arms: HIPEC
Drug: Adjuvant chemotherapy — Adjuvant chemotherapy using SOX or XELOX regimen will be administered as routine within 4-6 weeks.

SUMMARY:
The investigators intend to conduct a randomized controlled study to find if combining HIPEC (hyperthermic intraperitoneal perfusion chemotherapy) with post-neoadjuvant chemotherapy D2 resection could improve survival for patients with advanced gastric cancer, while comparing with the traditional approach of D2 resection after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Gastric cancer, as the second common malignant tumors in china, is marked by its poor prognosis and high recurrent rate. Although R0 resection could be achieved in most advanced gastric cancer(AGC) patients without metastasis, age-standardized 5-years survival rate was no more than 27.4%. Peritoneal metastasis accounts for 50% of the recurrent case and remain to be the most fatal recurrence pattern.

Hyperthermic intraperitoneal perfusion chemotherapy ( HIPEC ), has been proved as one of the most efficient approach against peritoneal carcinomatosis from gastric cancer and recommended in the guideline for gastric cancer published by the health committee of china. However, its role as prophylactic treatment after curative has never been determined. HIPEC works by delivering heat and cytotoxic drug to the cancer cell and is more effective on the tumor with small size. As present study suggest that Peritoneal metastasis is related to lymph node dissection during surgery while opening lymphatic channels and spreading viable cancer cells into the peritoneal cavity, HIPEC might be a reasonable approach to destroy the remaining cancer cells after curative surgery. Thus this research aim to explore the efficacy and safety of combining HIPEC (hyperthermic intraperitoneal perfusion chemotherapy) with post-neoadjuvant chemotherapy D2 resection.

ELIGIBILITY:
Inclusion Criteria:

1. First diagnosed as gastric cancer by pathological examination;
2. No previous chemotherapy or radiotherapy;
3. T stage:3-4, N stage: 1-3, M stage: 0, assessed by CT or ultrasound endoscope;
4. Eastern Cooperative Oncology Group performance status (ECOG PS): 0-1;
5. Informed consent signed;

Exclusion Criteria:

1. Other malignancy within 5 years.
2. Peritoneal metastasis detected during surgery.
3. Pregnant or lactating women;
4. Patients with conditions requiring emergency surgery;
5. Tumor progress during neo-adjuvant chemotherapy
6. Severe, uncontrolled physical or metal disease.
7. Poor compliance.
8. Uncontrolled infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of survival participants will be assessed according to the data collected by the followed up office. | 1-5 years

SECONDARY OUTCOMES:
Progression Free Survival | 1-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Sheng Peng, PhD, Principal Investigator — The sixth affliated hospital of Sun Yat-sen University
Locations (1):
- The sixth affliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marutsuka T, Shimada S, Shiomori K, Hayashi N, Yagi Y, Yamane T, Ogawa M. Mechanisms of peritoneal metastasis after operation for non-serosa-invasive gastric carcinoma: an ultrarapid detection system for intraperitoneal free cancer cells and a prophylactic strategy for peritoneal metastasis. Clin Cancer Res. 2003 Feb;9(2):678-85. PMID 12576435
- [Background] Lin CH, Hsieh HF, Yu JC, Chen TW, Yu CY, Hsieh CB. Peritoneal lavage with distilled water during liver resection in patients with spontaneously ruptured hepatocellular carcinomas. J Surg Oncol. 2006 Sep 1;94(3):255-6. doi: 10.1002/jso.20596. PMID 16900516
- [Result] Yonemura Y, de Aretxabala X, Fujimura T, Fushida S, Katayama K, Bandou E, Sugiyama K, Kawamura T, Kinoshita K, Endou Y, Sasaki T. Intraoperative chemohyperthermic peritoneal perfusion as an adjuvant to gastric cancer: final results of a randomized controlled study. Hepatogastroenterology. 2001 Nov-Dec;48(42):1776-82. PMID 11813623
- [Result] Hamazoe R, Maeta M, Kaibara N. Intraperitoneal thermochemotherapy for prevention of peritoneal recurrence of gastric cancer. Final results of a randomized controlled study. Cancer. 1994 Apr 15;73(8):2048-52. doi: 10.1002/1097-0142(19940415)73:83.0.co;2-q. PMID 8156509